CLINICAL TRIAL: NCT04739774
Title: Open-label, Non-randomized, One Sequence Cross-over Study to Investigate the Effect of Inhibition of CYP3A4/5 by Itraconazole on the Pharmacokinetics of CHF6001 in Healthy Subjects
Brief Title: Investigation of the Effect of Inhibition of CYP3A4/5 by Itraconazole on the PK of CHF6001 (Tanimilast)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CLI-06001AA1-11; 2020-003769-21 (EudraCT Number)
Record Dates: First submitted 2021-01-29; First posted 2021-02-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Itraconazole

STUDY DESIGN:
Intervention Model Description: one sequence cross-over design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment R (Experimental): Single dose of CHF6001
  Interventions: Drug: CHF6001 DPI
- Treatment T (Experimental): Single dose of CHF6001 administered after repeated doses of oral Itraconazole
  Interventions: Drug: CHF6001 DPI; Drug: Itraconazole

INTERVENTIONS:
Drug: CHF6001 DPI — Single dose of CHF6001
Drug: Itraconazole — Repeated doses of oral Itraconazole
  Arms: Treatment T

SUMMARY:
The objective of this proposed study is to investigate the pharmacokinetics interaction between CHF6001 as substrate and Itraconazole as inhibitor of CYP3A4/5 in a drug-drug interaction study.

DETAILED DESCRIPTION:
This clinical trial is a single centre, single dose Phase I study, with a non-randomized, open label, one sequence cross-over design.

A total of 24 healthy male and female are planned to be included.

Participants will be dosed with CHF6001 before and during co-administration of Itraconazole and will act as their own control. The study will be run with a one-sequence crossover design, where all subjects will be treated with CHF6001 in the first treatment period and CHF6001+Itraconazole in the second treatment period in order to avoid the need of a very long washout from the CYP3A4/5 inhibitor.

Standard safety assessments will be conducted during the Study, including safety blood and urine laboratory tests, vital signs, physical examinations, ECGs and observations of any adverse events. Blood samples will be also collected for PK analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's written informed consent obtained prior to any study-related procedure;
2. Healthy male and female subjects aged 18-55 years inclusive;
3. Ability to understand the study procedures, the risks involved and ability to be trained to use the inhalers correctly and to generate sufficient PIF using the In-Check device.
4. Body Mass Index (BMI) between 18,0 and 35,0 kg/m2 extremes inclusive;
5. Non- or ex-smokers who smoked < 5 pack years and stopped smoking > 1 year prior to screening;
6. Good physical and mental status
7. Vital signs within normal limits
8. 12 -lead digitalized Electrocardiogram (12-lead ECG) considered as normal
9. Pulmonary function test within normal limits
10. Women of Childbearing Potential (WOCBP) with fertile male partners: they and/or their partner must be willing to use a highly effective birth control method in addition to a barrier contraception method from the signature of the informed consent and until the follow-up visit. Males with non-pregnant WOCBP partners: they and or/ their partner must be willing to use a highly effective birth control method in addition to the male condom from the signature of the informed consent and until the follow-up visit. Males with pregnant WOCBP partner: they must be willing to use male contraception (condom) from the signature of the informed consent and until the follow-up visit

Exclusion Criteria:

1. Participation to another clinical trial where investigational drug was received, and last investigations were performed less than 8 weeks prior to screening;
2. Clinically relevant and uncontrolled respiratory, cardiac, hepatic, gastrointestinal, renal, endocrine, metabolic, neurologic, or psychiatric disorders, gastric surgery recent or in the past, and/or impaired gastric motility
3. Clinically relevant abnormal laboratory values
4. Abnormal liver enzymes at screening
5. Subjects with history of breathing problems
6. Positive HIV1 or HIV2 serology
7. Positive results from the Hepatitis serology
8. Blood donation or blood loss (equal or more than 450 ml) less than 2 months prior to screening or before the first dosing;
9. Positive urine test for cotinine
10. Documented history of alcohol abuse within 12 months prior to screening or a positive alcohol breath test
11. Documented history of drug abuse within 12 months prior to screening or a positive urine drug screen
12. Intake of non-permitted concomitant medications in the predefined period
13. Presence of any current infection, or previous infection that resolved less than 7 days prior to screening or before the first dosing;
14. Known intolerance and/or hypersensitivity to any of the excipients contained in the formulation used in the trial;
15. Known allergy to antifungal medicines;
16. Unsuitable veins for repeated venipuncture;
17. Heavy caffeine drinker
18. For females only: pregnant or lactating women. Serum pregnancy test to be performed at screening and urine pregnancy test to be performed before the first dosing;
19. Subjects receiving treatment with any drug known to have a well-defined potential for hepatotoxicity (e.g. isoniazide, nimesulide, ketoconazole) within the previous 3 months before the screening visit
20. Subjects using e-cigarettes within 6 months before screening.
21. Positive documented COVID-19 test before admission

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter (Cmax) | Over 96 hours after administration in blood
  Peak Plasma Concentration (Cmax) for CHF6001
Pharmacokinetic parameter (AUCt) | Over 96 hours after administration in blood
  Area under the plasma concentration versus time curve (AUCt) for CHF6001

SECONDARY OUTCOMES:
Pharmacokinetic parameter (AUC0-96) | Over 96 hours after administration in blood
  Area under plasma concentration from 0 to 96 hours (AUC0-96) for CHF6001, CHF5956 and CHF6095
Pharmacokinetic parameter (AUC0-∞) | Over 96 hours after administration in blood
  Area under curve extrapolated to infinity (AUC0-∞) for CHF6001, CHF5956 and CHF6095
Pharmacokinetic parameter (tmax) | Over 96 hours after administration in blood
  Time of the maximum plasma concentration (tmax) for CHF6001, CHF5956 and CHF6095
Pharmacokinetic parameter (t1/2) | Over 96 hours after administration in blood
  Terminal half-life (t1/2) for CHF6001, CHF5956 and CHF6095
Pharmacokinetic parameter (CL/F) | Over 96 hours after administration in blood
  Apparent systemic clearance (CL/F) for CHF6001
Pharmacokinetic parameter (AUCt) | Over 96 hours after administration in blood
  Area under the plasma concentration versus time curve (AUCt) for CHF5956 and CHF6095
Pharmacokinetic parameter (Cmax) | Over 96 hours after administration in blood
  Peak Plasma Concentration (Cmax) for CHF5956 and CHF6095

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Life Sciences - Clinical Pharmacology Unit Antwerpen, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No